CLINICAL TRIAL: NCT02610621
Title: IIT2015-11-Giuliano: Safety and Efficacy of Omission of Sentinel Node Biopsy for Breast Cancer Patients Who Plan to Have Adjuvant Chemotherapy
Brief Title: Safety and Efficacy of Sentinel Node Biopsy Omission for Breast Cancer Patients Who Plan to Have Adjuvant Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study may not be clinically relevant at this time.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Armando Giuliano, Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015-11-Giuliano-SNBO
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Clinically node negative; T1 and T2 invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lumpectomy without sentinel node biopsy (Experimental): Subjects will undergo standard of care lumpectomy. A biopsy of the sentinel node will not be performed. After surgery, subjects will receive standard of care radiation on the affected breast and chemotherapy.
  Interventions: Procedure: Lumpectomy without sentinel node biopsy

INTERVENTIONS:
Procedure: Lumpectomy without sentinel node biopsy — Biopsy of the sentinel node is considered standard of care treatment for women with localized breast cancer. The procedure will be eliminated at time of lumpectomy.

SUMMARY:
Eligible patients will be female, ages 18 and older and have a diagnosis of Clinical T1 or T2 invasive breast cancer with no suspicious palpable adenopathy. Patients will undergo standard of care lumpectomy without sentinel node biopsy and whole breast radiation, followed by chemotherapy.

Sentinel node biopsy is also considered standard care when patients have localized breast cancer. Treatment can often be influenced by whether the results of the biopsy show cancer or not. However, the biologic factors of the primary tumor have become more important in determining treatment recommendations in women with clinically node negative breast cancer.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the locoregional recurrence rate in patients with clinically node negative T1 and T2 breast cancer treated with systemic chemotherapy and whole breast irradiation in whom biopsy of the sentinel node is not performed. A locoregional recurrence is defined as any recurrence in the ipsilateral axillary nodes or in the supraclavicular nodes.

After surgery, a patient will receive standard of care radiation on her affected breast and chemotherapy. A physical examination of the affected breast and regional lymph nodes will be conducted every six months for the first two years of follow up and then yearly for the last 3 years of follow up. Imaging of the affected breast will occur every 12 months after surgery per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 and older, not pregnant or lactating
* Clinical T1 or T2 invasive cancer with no suspicious palpable adenopathy
* If abnormal axillary nodes are seen on preoperative imaging, a negative fine needle aspiration or core biopsy is required for study entry.
* Planned treatment with breast conserving surgery and whole breast irradiation
* Chemotherapy required postoperatively based on patient and tumor characteristics at diagnosis

Exclusion Criteria:

* Patients with suspicious palpable axillary adenopathy
* Patients with biopsy demonstrating axillary nodal metastases
* Patients with treatment by mastectomy
* Patients who have undergone neoadjuvant chemotherapy
* Patients with co-morbidities rendering the patient not a candidate for chemotherapy, surgery, or irradiation
* Patients treated with accelerated partial breast irradiation (APBI)
* Patients with contraindication to radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
A determination of the locoregional recurrence rate in patients with clinically node negative T1 and T2 breast cancer treated with systematic chemotherapy and whole breast radiation in whom sentinel node biopsy is not performed | Assessed up to 5 years from date of lumpectomy

CONTACTS AND LOCATIONS:
Overall Officials: Armando Giuliano, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States